CLINICAL TRIAL: NCT03753516
Title: Pelvic Floor Support After Laparoscopic Hysterectomy for Benign Conditions: A Randomized Controlled Trial Comparing Vaginal Cuff Closure Techniques
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with follow up 2/2 COVID-19 Pandemic
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRNMMC-2017-0055
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic - Vaginal Cuff Closure (Active Comparator)
  Interventions: Procedure: Laparoscopic - Vaginal Cuff Closure
- Vaginal - Vaginal Cuff Closure (Active Comparator)
  Interventions: Procedure: Vaginal- Vaginal Cuff Closure

INTERVENTIONS:
Procedure: Laparoscopic - Vaginal Cuff Closure — All participants are scheduled for either laparoscopic or robotic assisted total hysterectomy. At the end of the hysterectomy the vaginal cuff is closed. In this arm the vaginal cuff will be close laparoscopically using an 0-Barbed suture.
  Arms: Laparoscopic - Vaginal Cuff Closure
Procedure: Vaginal- Vaginal Cuff Closure — All participants are scheduled for either laparoscopic or robotic assisted total hysterectomy. At the end of the hysterectomy the vaginal cuff is closed. In this arm the vaginal cuff will be close vaginally using an 0-Vicryl suture in a vertical fashion.
  Arms: Vaginal - Vaginal Cuff Closure

SUMMARY:
The purpose of this study is to learn about the effect of different vaginal cuff closure techniques on pelvic support after laparoscopic hysterectomy and robotic assisted laparoscopic hysterectomy for benign gynecologic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age undergoing total laparoscopic hysterectomy and robotic assisted total laparoscopic hysterectomy for benign disease.
* Subjects must be able to self-consent.
* Department of Defense beneficiary

Exclusion Criteria:

* Patients will be excluded if they undergo a concurrent procedure for prolapse.
* If the indication for the procedure is a malignancy.
* Those that plan to leave the area in less than 1 year will not be included.
* Pop-Q Point C of >-4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse - Quantification Point C | 6-8 weeks post op
  The Pelvic Organ Prolapse - Quantification system is a validated way to measure pelvic organ prolapse. The investigators will measure this post op at 6-8 weeks to see if prolapse is better using one method vs the other.
Pelvic Organ Prolapse - Quantification Point C | 1 year post op
  The Pelvic Organ Prolapse - Quantification system is a validated way to measure pelvic organ prolapse. The investigators will measure this post op at 1 year to see if prolapse is better using one method vs the other.

SECONDARY OUTCOMES:
Vaginal Cuff Dehiscence | 1 year
Vaginal Cuff Abscess | 1 year
Vaginal Cuff Cellulitis | 1 year
Vaginal Cuff bleeding | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No